CLINICAL TRIAL: NCT05750693
Title: Impact of Somatic PIK3CA Mutations on Pathological Complete Response (pCR) in HER2-positive Early Breast Cancer.
Brief Title: PIK3CA in HER2+ BC and pCR Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4469
Record Dates: First submitted 2023-02-20; First posted 2023-03-02 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-02

CONDITIONS: HER2-positive Breast Cancer
Keywords: PIK3CA; Neoadjuvant chemotherapy; pathologic complete response; Her-2
MeSH Terms: conditions — Hereditary Sensory and Autonomic Neuropathies; Pathologic Complete Response

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients who received neoadjuvant chemotherapy (Experimental): Breast cancer samples of paraffin embedded tissue, obtained from the waste material of the diagnostic core-biopsy, stored at the Pathological Anatomy Service, will be used in order to analyze PIK3CA mutations status.
  Interventions: Genetic: PIK3CA analysis

INTERVENTIONS:
Genetic: PIK3CA analysis — PIK3CA will be investigated together with HER2 in pre-NAD tissue samples, in order to evaluate the correlation with response to NAD chemotherapy, with a 16-gene MYRIAPOD kit. This evaluation will be performed on all 58 patients in the study for group (responders and not responders).
  Moreover 10 patient samples (5 responders and 5 non-responders) will be subjected to gene expression profile analysis. Specifically, a transcriptomic analysis will be performed on total RNA from one inch of cells (10-50 cells isolated by LCM from FFPE biopsy, RNA seq) which will allow to have the transcriptional profile for each patient of protein-coding transcripts (coding RNAs) and long non-coding RNAs.
  In addition, an NGS analysis by TSO500 will be performed in parallel, on the slide following the previous one, to have the genome sequence (523 genes) on the same 10-50 cells isolated by LCM from FFPE biopsy for the identification of any mutations.

SUMMARY:
The goal of the study is to evaluate the impact of somatic PI3KCA mutations on pCR in HER2-positive early breast cancer in real life. The main question it aims to answer iS.

- Is there a correlation between PIK3CA mutations and response to neoadjuvant chemotherapy in HER2 early breast cancer? Participants who received neoadjuvant chemotherapy in addition to anti-Her2 target therapy will undergo PIK3CA analysis in order to answer to this question.

DETAILED DESCRIPTION:
Women with breast cancer (BC) overexpressing HER2 have more aggressive tumors and, without administration of anti-HER2agents, a shorter disease-free survival (DFS) and overall survival (OS) compared to patients with HER2-negative subtypes. Since the introduction of trastuzumab, the course of HER2-positive BC has notably improved in both metastatic and early settings. Indeed, anti-HER2 treatment has influenced the response to neoadjuvant (NAD). Women with breast cancer (BC) overexpressing HER2 have more aggressive tumors and, without administration of anti-HER2agents, a shorter disease-free survival (DFS) and overall survival (OS) compared to patients with HER2-negative subtypes. Since the introduction of trastuzumab, the course of HER2-positive BC has notably improved in both metastatic and early settings. Indeed, anti-HER2 treatment has influenced the response to neoadjuvant (NAD) therapy in HER2-positive BC by increasing the pCR rate. However, primary and acquired resistance to trastuzumab-containing regimens remains one of the major issues in clinical practice. Selecting patients that will benefit from anti-HER2 treatment is therefore essential. Overexpression of HER2 is identified in ∼20% of early-stage invasive BC and induces the downstream activation of the PI3K/AKT/mTOR pathway that plays a crucial role in developing resistance to trastuzumab: PIK3CA mutation and PTEN protein loss cause an hyperactivation of the pathway, whereas PIK3CA wild-type and retained or increased PTEN expression lead to a lower activation. PIK3CA mutations are predominantly found in hotspots located in the helical and kinase domains (exons 9 and 20), resulting in activation of the kinase. Another potential mechanism of resistance to trastuzumab is the estrogen receptor (ER) in those tumors that express both ER and HER2. To date, resistance biomarkers are lacking: despite the fact that data on PIK3CA mutations demonstrate significantly lower pCR rates, this has not led to an inclusion of the marker into routine diagnostics. PIK3CA can be investigated together with HER2 in pre-NAD tissue samples, in order to evaluate the correlation with response to NAD chemotherapy. That is an optimal setting to understand if PI3K could be considered a biomarker for HER2 therapy-resistant tumors and to select patients with poorer prognosis.

This study investigates the association of pCR with PIK3CA mutations and ER status and their prognostic value in HER2-positive BC treated with anti-HER2 therapy in addition to NAD chemotherapy.

Response to NAD therapy will be determined as pCR, defined as no invasive residuals in breast tissue and lymph nodes (ypT0/is, ypN0). Disease-free survival (DFS) will be defined as time in months from randomization to (local or distant) disease recurrence, secondary malignancy or death due to any cause. Overall survival (OS) was defined as time in months from randomization to death due to any cause.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent.
* Age older than 18 years.
* Unilateral or bilateral primary carcinoma of the breast, confirmed histologically by core biopsy.
* Tumor lesion in the breast with a palpable size of ≥ 2 cm and/or ≥ 1.5 cm by ultrasound or magnetic resonance imaging (MRI). In case of inflammatory carcinoma the extent of inflammation can be used as measurable lesion.
* American Joint Commission on Cancer stage II or III invasive breast cancer.
* Known estrogen (ER)- and progesterone (PgR)-receptor negative or positive tumors.
* Known HER-2/neu positive tumors, defined as HercepTest IHC 3+ or SISH+.
* Patients suitable for neoadjuvant chemotherapy
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) ≤2 or Karnowsky performance status index at least 80%.
* Normal cardiac function must be confirmed by ECG and cardiac ultrasound (LVEF or shortening fraction) within 1 month prior to registration.
* Laboratory requirements:

  * Hematology: Absolute neutrophil count (ANC) ≥ 1.5 x 109/L, platelets ≥ 100 x 109/L, Hemoglobin ≥ 10 g/dL.
  * Hepatic function: Total bilirubin < 1 x UNL, ASAT (SGOT) and ALAT (SGPT)≤ 2.5 x UNL, Alkaline phosphatase ≤ 5 UNL. Patients with ASAT and / or ALAT > 1.5 x UNL associated with alkaline phosphatase > 2.5 x UNL are not eligible for the study.
  * Renal function: Creatinine ≤ 2 mg/dL, < 1,25 UNL (or the calculated creatinine clearance ≥ 60 mL/min).
  * Paraffin tumor tissue block made available.
  * Availability to provide the set up of the histological preparations for molecular analysis.
  * Negative pregnancy test (urine or serum).
  * Patients must be available and compliant for treatment and follow-up.

Exclusion Criteria:

* Patients candidate for adjuvant chemotherapy.
* Evidence of distant metastasis.
* Prior chemotherapy for any malignancy.
* Prior radiation therapy for breast cancer.
* Pregnant or lactating patients.
* Inadequate general condition.
* Previous malignant disease.
* Known or suspected congestive heart failure (>NYHA I) and/or coronary heart disease, angina pectoris requiring antianginal medication, previous history of myocardial infarction, evidence of transmural infarction on ECG, un- or poorly controlled arterial hypertension, rhythm abnormalities requiring permanent treatment, clinically significant valvular heart disease.
* History of significant neurological or psychiatric disorders that would prohibit the understanding and giving of informed consent.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2022-05-02 (Actual); Primary Completion 2023-09-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
pathologic complete response | 7 months
  To investigate the association of pCR and PIK3CA mutations in patients with locally advanced HER-2 positive Breast Cancer.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Rome, RM, Italy

IPD SHARING:
Plan to Share IPD: No